CLINICAL TRIAL: NCT05322382
Title: Accuracy of Pulse Oximeters With Profound Hypoxia - Test Protocol
Brief Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 008_SPO_CV_OS_USF
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: SpO2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Subjects undergo an interventional procedure and non-invasive measurements of SpO2.
  Interventions: Procedure: A-line

INTERVENTIONS:
Procedure: A-line — Subjects breathe air mixtures containing reduced amounts of oxygen to produce the desired level of hypoxemia.
  Other Names: Hypoxemia

SUMMARY:
This project aims to test the accuracy of pulse oximeters during mild, moderate, and severe hypoxia, i.e., a range of arterial HbO2 saturation from 100 down to 70%. A typical study will include at least ten subjects (at least 200 necessary data points to meet the ISO 80601-2-61:2017).

DETAILED DESCRIPTION:
After local anesthetic injection, a 22-gauge catheter is inserted in one radial artery. Pulse oximeters are attached to fingers, ears, or flat body surfaces. Subjects are in a comfortable semi-recumbent position. Subjects then breathe air mixtures containing reduced amounts of oxygen to produce the desired level of hypoxemia. Stable, safe, and controlled hypoxia is breath-by-breath by breath respiratory gas analysis and a computer program that permits the inspired gas mixture to be adjusted to achieve a level of lung alveolar gas that will achieve the desired degree of saturation.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>30).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. Subject has diabetes.
5. Subject has a clotting disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of pulse oximeter with profound hypoxia | 2 days
  Perform accurate measurement of a range of arterial HbO2 saturation from 100 to down to 70% during mild, moderate, and severe hypoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, Principal Investigator — UCSF Hypoxia Lab
Locations (1):
- University of California at San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No